CLINICAL TRIAL: NCT06929221
Title: The Effect of Bedside Whiteboard Use on Anxiety, Depression and Nursing Care in Chronic Obstructive Pulmonary Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Agri Ibrahim Cecen University (Other)
Responsible Party: Principal Investigator, Ramazan DENİZ, Principal Investigator, Agri Ibrahim Cecen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RDENİZ02
Record Dates: First submitted 2025-03-22; First posted 2025-04-16 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-04

CONDITIONS: COPD; Nursing Care
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Whiteboard group (Experimental)
  Interventions: Other: use of whiteboard
- Control Group (No Intervention)

INTERVENTIONS:
Other: use of whiteboard — Patients will be followed up for 7 days. Routine nursing care will be applied to the control group. The following information will be included on the whiteboard fixed in the patient room for the intervention group.
  * Nurse's name
  * Doctor's name
  * Treatment times during the day
  * Nursing interventions and hours for the diagnoses considered for the patient's major problems
  * Timing of diagnostic and imaging techniques to be performed on the patient
  * Content of appropriate discharge education for the patient
  * Points to be considered by the patient before and after treatment
  * Dietary considerations for the patient
  * Nurse and patient's private note As a result of the data obtained, statistical analyses will be performed and interpreted to determine the effect of whiteboard use on anxiety, depression and satisfaction with nursing care in COPD patients.
  Arms: Whiteboard group

SUMMARY:
ABSTRACT Chronic obstructive pulmonary disease (COPD) is a disease characterized by the inability of the body to adequately exchange gases, resulting in progressive shortness of breath that can form secretions and compromise the performance of daily activities. COPD is reported as the third most common cause of death worldwide, with 3.23 million deaths in 2019. Anxiety and depression are common in individuals with COPD. However, COPD is more common in patients with other chronic diseases such as hypertension, diabetes, cancer or musculoskeletal disorders. Communication is a key component in interprofessional care as well as in improving patient care outcomes. Strategies to address gaps in the quality of information and communication between patients, caregivers and professionals improve patient safety as well as quality of care. One of these strategies is the use of whiteboards at the bedside. The use of whiteboards at the bedside has emerged as a strategy to improve interprofessional team participation, communication and information sharing with care teams, patients and families. This study will be conducted in randomized controlled single blind parallel groups to examine the effect of bedside whiteboard use on anxiety, depression and nursing care satisfaction in COPD patients. The research will consist of patients who are hospitalized in Atatürk University Research Hospital Chest Diseases Clinic and who meet the inclusion criteria. In the results of the research, it is thought that the use of whiteboard will affect the communication between health care team members.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Having a medical diagnosis of COPD
* To be in a condition to be followed up with at least 7 days

Exclusion Criteria:

* - Having strong reading and comprehension skills

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
How does the use of whiteboard affect anxiety, depression and nursing care satisfaction in COPD patients? | From registration until the end of the 3th month
  The Hospital Anxiety and Depression Scale will be used to examine the effect of the whiteboard to be used for COPD patients on anxiety and depression. A total scale score of 28 and above indicates a high level of anxiety and depression.
How does the use of whiteboard affect anxiety, depression and nursing care satisfaction in COPD patients? | From registration until the end of the 3th month
  The Patient Satisfaction with Nursing Care Quality Questionnaire Scale will be used to examine the effect of the whiteboard to be used for COPD patients on nursing satisfaction. A total score of 47.5 and above indicates high nursing care satisfaction.